CLINICAL TRIAL: NCT06691308
Title: Clinical Study Evaluating the Safety and Efficacy of WL276 CAR-T Cell Therapy in CD276 Positive Recurrent or Progressive Glioblastoma Patients
Brief Title: WL276 CAR-T Cell Therapy for CD276 Positive Recurrent or Progressive Glioblastoma Patients
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WL276001
Record Dates: First submitted 2024-11-05; First posted 2024-11-15 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Recurrent or Progressive Glioblastoma
Keywords: WL276 CAR-T cells; CD276 positive
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD276 positive recurrent or progressive glioblastoma (Experimental): Inject WL276 CAR-T cells through local intracranial administration using the Ommaya device, once a week for 3 weeks. After 3 weeks of continuous administration, perform cranial MRI imaging to evaluate tumor progression and assess drug efficacy. Propose to deliver doses of 5 * 10 ^ 6 CAR-T Cells and 1 * 10 ^ 7 CAR-T Cells in sequence, with 3 subjects enrolled in each dose group
  Interventions: Combination Product: WL276 CAR-T cells

INTERVENTIONS:
Combination Product: WL276 CAR-T cells — This study intends to include 6 subjects, with 3 subjects receiving 5 * 10 ^ 6 CAR-T Cells and 3 subjects receiving 1 * 10 ^ 7 CAR-T Cells at different doses

SUMMARY:
Clinical study evaluating the safety and efficacy of WL276 CAR-T cell therapy in CD276 positive recurrent or progressive glioblastoma patients

DETAILED DESCRIPTION:
This study is an open label, single center early exploratory clinical trial of WL276001 CAR-T cell therapy for CD276 positive recurrent or progressive glioblastoma patients. This study used an improved "3+3" experimental design for dose escalation to explore the safety and efficacy of in-situ administration of WL276001 CAR-T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with glioblastoma through histopathological examination;
2. Patients with unresectable recurrent or progressive glioblastoma who have failed or are intolerant to standard treatment; 8.1The standardized systematic treatment received by patients must comply with the 2022 edition of the "Guidelines for the Treatment of Gliomas"; 8.2Requirements for treating intolerance: Refers to patients who are unable to continue the current effective systemic standardized treatment due to toxic side effects such as vomiting, diarrhea, abdominal pain, bone marrow suppression, etc. of grade ≥ 3. Refusal due to economic or personal reasons is not accepted;
3. Age ≥ 18 years old, including boundary values;
4. Expected survival period greater than 2 months;
5. There is at least one measurable intracranial lesion that meets the criteria of Neuro Tumor Response Evaluation (RANO);
6. Patients must provide tumor samples within 2 years that meet the requirements (paraffin blocks or unstained sections with a quantity that meets the testing requirements specified in this study) and have positive CD276 expression detected by immunohistochemistry;
7. Karnofsky (KPS) functional status score ≥ 60 points;
8. Blood routine:

   8.1Hemoglobin (Hb) ≥ 90g/L; 8.2Absolute neutrophil count (ANC) ≥ 1.5 × 10 ^ 9/L; 8.3Platelet count (PLT) ≥ 70 × 10 ^ 9/L; 8.4Absolute value of lymphocytes ≥ 0.5 × 10 ^ 9/L;
9. The liver, kidney, heart, and lung functions meet the following requirements:

   9.1Creatinine clearance rate ≥ 60ml/min; 9.2Alanine transaminase (ALT) and aspartate transaminase 9.3Aspartate aminotransferase (AST) ≤ 2.5 × ULN, total bilirubin (TBL) ≤ 1.5 × ULN (for the elevation of ALT and AST that can be explained by liver invasion, AST and ALT high limit can be upregulated up to 5-fold, and TBL high limit can be upregulated up to 3-fold); 9.4Serum albumin ≥ 3.0g/dL; 9.5Left ventricular ejection fraction ≥ 50%, no pericardial effusion [ECHO (Echocardiography, ECHO) examination], no clinically significant ECG (Electrocardiogram, ECG) results; 9.6Blood oxygen saturation is greater than 95% under non oxygen inhalation conditions.
10. Women of childbearing age who have a negative blood pregnancy test before the start of the trial and agree to take effective contraceptive measures during the trial period until the last follow-up; Male participants with reproductive partners agree to take effective contraceptive measures during the trial period until the last follow-up;
11. Those who voluntarily participate in this experiment and sign the informed consent form.

Exclusion Criteria:

1. Those who require the use of immunosuppressants; Or individuals with autoimmune diseases;
2. Patients who have received or are waiting for organ transplantation in the past;
3. The toxicity caused by previous treatment has not stabilized or recovered to ≤ level 1 (except for cases judged by the researcher to be clinically insignificant);
4. There is a large amount of uncontrollable serosal fluid accumulation (such as pleural effusion, abdominal effusion, pericardial effusion) after treatment;
5. Use any of the following drugs or treatment methods within the specified time before cell collection:

   5.1Used therapeutic doses of corticosteroids within one week prior to cell collection. But the use of topical and inhaled steroids is allowed; 5.2Received chemotherapy drugs within one week prior to cell collection. If the oral chemotherapy drug has passed at least 3 half lives before cell collection, it is allowed to be included in the group; 5.3Individuals who use drugs to stimulate bone marrow hematopoietic cell production within 5 days prior to cell collection;
6. CNS diseases that have clinical significance in the past or screening, and have been assessed by researchers as having safety risks;
7. Individuals who have previously used any gene therapy products;
8. Active hepatitis B or hepatitis C virus is defined as: subjects who are positive for hepatitis B B virus surface antigen (HBsAg) or hepatitis B B core antibody (HBcAb) and whose peripheral blood HBV DNA titer is higher than the upper limit of detection; Individuals with positive hepatitis C virus (HCV) antibodies and positive peripheral blood HCV RNA (HCV RNA); People infected with AIDS virus and syphilis;
9. Active EBV and cytomegalovirus are defined as patients with positive or negative IgM antibodies in EBV serum but EBV-DNA levels higher than normal; Patients with IgM antibody positive or IgM antibody negative but CMV-DNA higher than normal in the serum of cytomegalovirus (CMV);
10. Used the research drug within 4 weeks prior to cell collection. But if the experimental treatment is ineffective or if the disease progresses, and at least 5 half lives have passed before cell collection, it is allowed to be included in the group;
11. Received radiation therapy within 4 weeks prior to cell collection;
12. Patients who have undergone major surgical procedures or significant trauma within 4 weeks prior to cell collection, or who are expected to undergo major surgery during the study period;
13. If immunotherapy such as anti-PD1 and PD-L1 has been used before cell infusion, at least 5 half lives must be passed between the last dose and CAR-T cell infusion;
14. Abnormal cardiac function includes: long QTc syndrome or QTc interval>480 ms; Complete left bundle branch block, grade II/III atrioventricular block; Severe and uncontrolled arrhythmias requiring medication treatment; History of chronic congestive heart failure and NYHA ≥ 3 (refer to Appendix 4) with a heart ejection fraction below 50% within the 6 months prior to screening; Heart valve disease with CTCAE ≥ 3 grade; Within the first 6 months of screening, there has been a history of myocardial infarction, cardiac angioplasty or stent implantation, unstable angina, severe pericardial disease, or other clinically significant heart diseases;
15. Patients who require anticoagulant therapy;
16. Patients requiring long-term antiplatelet therapy;
17. Start screening for symptomatic history of venous thrombosis or pulmonary embolism within the previous 6 months;
18. History of malignant tumors other than non melanoma skin cancer or carcinoma in situ (such as cervical, bladder, breast) (unless in a disease-free state for at least 3 years);
19. Infections (fungal, bacterial, viral, or other) that require intravenous injection of antibiotics for control or are uncontrollable, such as simple urinary tract infections and bacterial pharyngitis, can be included if the researcher evaluates that they can be controlled through treatment;
20. Unable to perform MRI examination (such as installing pacemakers, metal dentures, etc.)
21. The researcher shall determine whether the patient has any factors that affect compliance with the protocol, or is unwilling or unable to comply with the procedures required in the research protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-11-12 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety（Adverse event incidence rate、Incidence rate of abnormal laboratory test results） and tolerability（DLT incidence rate） of WL276 CAR-T cell therapy for CD276 positive recurrent or progressive glioblastoma | Within 28 days after infusion
  Adverse events related to CAR-T cell therapy within 28 days after infusion, abnormal laboratory test results with clinical significance, including dose limiting toxicity (DLTs).

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 720 days after infusion
  Progression Free Survival (PFS) after infusion.
Overall Survival (OS) | 720 days after infusion
  Overall Survival (OS) after infusion.

OTHER OUTCOMES:
incidence of adverse events | 720 days after infusion
  Collect and compare the safety (incidence of adverse events) of different administration methods
disease improvement rate | 720 days after infusion
  Collect and compare the efficacy (disease improvement rate) of different administration methods
CAR-T cell counting | 720 days after infusion
  Collect and compare cell expansion data (CAR-T cell counts) after different administration methods
CAR-T cell survival rate | 720 days after infusion
  Retention of WL276 CAR-T cells in peripheral blood, cerebrospinal fluid, and/or tumor tissue of patients
CAR-T cell survival time | 720 days after infusion
  Duration of WL276 CAR-T cells in peripheral blood, cerebrospinal fluid, and/or tumor tissue of patients
Cytokine levels | 720 days after infusion
  Changes in cytokines in peripheral blood of subjects before and after infusion of WL276 CAR-T cells, as well as the time to return to normal

CONTACTS AND LOCATIONS:
Overall Officials: gang Cheng, doctorate, Principal Investigator — Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: No